CLINICAL TRIAL: NCT06236256
Title: Advanced Hybrid Closed Loop System (780G) for People With Type 1 Diabetes Mellitus Patients Over the Age of 60: Efficacy in Improving Glucose Indices, Quality of Life, Cognitive Functions and Physical Capacity
Brief Title: Advanced Hybrid Closed Loop System (AHCL) in Older Patients With Type 1 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Tali Cukierman-Yaffe, Professor, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0205-23-SMC
Record Dates: First submitted 2023-11-14; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Older; Physical capacity; Frailty; Cognitive function
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Frailty | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AHCL group (Experimental): Participants will be connected to the MiniMed 780G AHCL system for the 12 months study period. This group will have two additional visits to allow for patients to be trained on the AHCL system.
  Interventions: Device: MiniMed™ 780G Advanced Hybrid Closed Loop (AHCL) system
- MDI/CSII group (Placebo Comparator): The patient will continue MDI/CSII treatment as per their routine procedures. At the beginning, middle and end of the stage they will be connected to a standalone sensor from which glucose data will be collected.
  Interventions: Other: MDI/CSII

INTERVENTIONS:
Device: MiniMed™ 780G Advanced Hybrid Closed Loop (AHCL) system — The MiniMed™ 780G Advanced Hybrid Closed Loop (AHCL) system consists of the following devices: MiniMed 780G insulin pump, Guardian Link (4) transmitter and the Guardian Sensor (4). It is intended for continuous delivery of basal insulin at selectable rates, and the administration of insulin boluses at selectable amounts for the management of type 1 diabetes mellitus. The system is also intended to continuously monitor glucose values in the fluid under the skin. The MiniMed 780G system includes SmartGuard technology, which can be programmed to automatically adjust insulin delivery based on continuous glucose monitoring (CGM) sensor glucose values and can suspend delivery of insulin when the SG value falls below or is predicted to fall below predefined threshold values. Study participants will be connected to the system and glucose data will be collected throughout the 12 month study period.
  Arms: AHCL group
Other: MDI/CSII — Participants in the control group with continue their routine procedures that include eighter Multiple daily insulin injections (MDI) treatment or different kinds of Continuous subcutaneous insulin infusion (CSII) pumps depending on their treatment before the study. The participants will be connected to a standalone sensor at the start, middle and end of the study and glucose data will be collected.
  Arms: MDI/CSII group

SUMMARY:
The trial is a randomized controlled, parallel group design study. Patients will be followed up during approximatively 12 months.

Patients will be randomized to either the MDI/CSII group which will continue their treatment as per routine procedures and the advanced Hybrid Closed Loop system (AHCL) group which will be connected to the Minimed 780G system. .

At the end of the 12 month study period, we will evaluate whether the AHCL system improved glucose indices in older individuals with Type 1 diabetes mellitus (T1DM) and assess whether the ACHL treatment improved physical capacity, frailty & sarcopenia indices as well as quality of life and cognitive functions.

DETAILED DESCRIPTION:
All participants will go through a screening phase that includes an eligibility assessment, informed consent forms, Cognitive function assessment ( QoL questionnaire, WHO-5 questionnaire, MOCA, DSST, General Heath question), Sarcopenia/functional status/frailty assessment ( Timed up and Go , 6 min walk, 10 meter walk, Berg Balance Scale , Four Square Step Test , Grip Strength, 30 second chair stand, Fried Scale) and Lab tests.

After the screening, the participants will start a two week run in phase while continuing their routine procedures with an added unblinded G4 guardian standalone sensor.

sensor and data will be collected for 14 days and afterwards patients will be randomized to either the MDI/CSII group which will continue their treatment as per routine procedures and the AHCL group which will be connected to the Minimed 780G system. Both groups will have a similar number of visits in order to minimize bias. However, the AHCL group will have 2 additional visits to allow for patients to be trained on the AHCL system. After 6 months, both groups will be connected to the standalone sensor and glucose data will be collected after 2 weeks.

After 12 months of the study period, all participants will undergo primary assessments, blood tests questionnaires and will finish their part in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 60 years
2. T1DM
3. Willing to participate in a study for the specified duration
4. Willing to perform ≥ 4 finger stick blood glucose measurements daily or connected to a "basket approved" CGM
5. Willing to wear the system continuously throughout the study
6. Treated with MDI/CSII (with exclusion of 780G or other hybrid closed systems)
7. Lack of advanced complications of diabetes

Exclusion Criteria:

1. Severe concurrent illness
2. Laboratory abnormalities, or medications that might affect study participation,
3. Severe renal impairment
4. Any illness that may interfere with study procedures

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Improvement of glucose measures in older individuals | 12 months
  The primary objective of this study is to evaluate whether the AHCL (MiniMed 780G) system improves glucose indices in older (above 60 years of age) individuals with Type 1 diabetes mellitus.
  Glucose differences between the groups will be monitored and evaluated by difference in the percentage of time spent within range with sensor glucose (SG) between 70-180 mg/dL (Primary outcome), time in hyperglycemic range SG > 250 mg/dL , SG > 180 mg/dL, time in hypoglycemic range with SG < 70 mg/dL , SG < 54 mg/dL as well as difference in the glycemic variability, mean glucose level and change in HbA1c levels.

SECONDARY OUTCOMES:
Time up and go | 12 months
  The test measures the ability of a person to: stand up, walk, turn around and sit down safely in a timely manner. The test examines most mobility skills. The participant is told to get up from a chair with handles, walks 3 meters, turns, walks back, and sit down again. The score is according to the length of time in seconds to complete the task. The score is categorized according to the risk for falls and independent walking. The following cut-offs are conventionally used: less than14 seconds = independent mobility; 15-20 seconds= semi-independent mobility may have a some what increased risk for falls & needs further evaluation some may need a walking aid; 20-30 seconds= dependent mobility: need help walking, 50% with a cane, 40% walker, 10% supervision. Some will need help in transfers, and most will require help using the toilet.
6 minute walk | 12 months
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. The six minute walk distance in healthy adults has been reported to range from 400m to 700m. People with lower vs. higher scores on the 6 minute walk are at higher risk for falls, disability, frailty, hospitalization and death. There is no conventional cut offs, however as with other tests, severe impairment may be defined as two standard deviations below the norm.
Four Square Step Test (FSST) | 12 months
  The Four Square Step Test (FSST) evaluates dynamic balance in a high functional level and features walk forward backwards left and right above two, 90 cm and 2.5 cm high long sticks that divide the floor into four squares. The participant is stands in square 1 facing no. 2 square. The goal is to walk as quickly as possible in all the squares in the following order: from 1 to- 2,3,4,1,4,3,2 and 1 without touching the sticks. The score is the time required to complete the entire route. Sever physical impairment is considered less then 15 seconds, Mild physical impairment is considered 10.14- 14.59 seconds, intact physical impairment is considered less then 10.14 seconds.
Grip strength | 12 months
  The maximum grip strength is examined utilizing the Jammer dynamometer. The test is conducted in a neutral hand position and repeated three times. The score is the average strength in kg this is compared to the general population according to age and gender. There is no conventional cut offs, however as with other tests, severe impairment may be defined as two standard deviations below the norm.

OTHER OUTCOMES:
Fried scale | 12 months
  Fried scale criteria is used for identifying frailty in older people. Frailty is defined as the presence of at list three components. i. Weight loss: More then 10 pounds unintentional weight loss in the past year (not due to dieting or exercise).
  ii. Poor endurance and energy: as indicated by self-report of exhaustion. Self-report exhaustion, identified by two questions from the CES-D scale.
  iii. Low Physical Activity level: kilocalories expended per week, calculated adjusted according to age and gender.
  iv. Walk time: over seven seconds to pass three meters
Moca | 12 months
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MOCA), a rapid screening tool for mild cognitive dysfunction. It assesses different cognitive domains such as: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. A MoCa score<21 was defined as severe cognitive impairment (probable dementia). A MoCA score between 21-25 was defined as mild cognitive impairment.
DSS | 12 months
  The Digit Symbol Substitution Test (DSST): a subtest of the Wechsler Adult Intelligence Scale (3rd Edition) and pertains to a wide array of cognitive domains such as visual-motor speed and coordination, capacity for learning, attention, concentration and short term memory. The DSST gets a raw score between 0 and 90 which can then be converted to a standardized score with a mean score of 10 and a standard deviation of 3.
WHO-5 | 12 months
  The WHO-5 wellbeing questionnaire asses emotional status. Who 5 gets a raw score of 0 to 25 which is then multiplied by 4 to convert the score to a continuum between 0 (worst imaginable quality of life) to 100 (best imaginable quality of life). A score of ≤50 indicates poor wellbeing and suggests further investigation into possible symptoms of depression. A score of 28 or below is indicative of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba medical center, Ramat Gan, Israel